CLINICAL TRIAL: NCT00641095
Title: Phase III, Multicentre, Randomised Study of Fludarabine/Cyclophosphamide Combination With or Without Rituximab in Patients With Untreated Mantle Cell Lymphoma
Acronym: MCLPIII
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/06/052; 2006-001965-41 (EudraCT Number); MREC-02/6/31 (Other: South West Multi-centre Research Ethics Committee); ISRCTN (Registry Identifier: NCT00641095)
Record Dates: First submitted 2008-03-20; First posted 2008-03-21 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fludarabine/Cyclophosphamide/Rituximab (Experimental): Fludarabine 40mgs/m2 oral days 1-3 Cyclophosphamide 250mgs/m2 oral days 1-3 Rituximab 375mgs/m2 day 1 iv infusion
  Every 28 days
  Interventions: Biological: rituximab; Drug: Cyclophosphamide; Drug: Fludarabine
- Fludarabine/Cyclophosphamide (Active Comparator): Fludarabine 40mgs/m2 oral days 1-3 Cyclophosphamide 250mgs/m2 oral days 1-3
  Every 28 days
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: rituximab — concentrate for solution for infusion
  Arms: Fludarabine/Cyclophosphamide/Rituximab
Drug: Cyclophosphamide — Tablets
Drug: Fludarabine — Film coated tablet

SUMMARY:
This randomized phase III trial is comparing how well fludarabine and cyclophosphamide work when given together with or without rituximab in treating patients with previously untreated mantle cell lymphoma.

DETAILED DESCRIPTION:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. It is not yet known whether giving combination chemotherapy together with rituximab is more effective than combination chemotherapy alone in treating mantle cell lymphoma.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine phosphate IV or orally once daily and oral cyclophosphamide once daily on days 1-3. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive rituximab IV on day 1 and fludarabine phosphate IV or orally once daily and oral cyclophosphamide once daily on days 1-3. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow and blood sample collection periodically for molecular studies. Samples are analyzed for morphology; sIgM, sIgD, CD19, CD20, CD5, CD10, CD23, bcl-1, bcl-6 via immunophenotyping and immunohistochemistry; and t(11,14) translocation via interphase fluorescence in situ hybridization (FISH) mutational analysis.

After completion of study treatment, patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

This trial follows on from the Phase II randomised study of fludarabine/cyclophosphamide combination with or without Rituximab in patients with untreated mantle cell lymphoma. ISRCTN number: NCT00053092

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mantle cell lymphoma (MCL), meeting the following criteria:

  * Diagnosis confirmed by examination of representative material (lymph nodes or bone marrow) together with a typical immunophenotype CD5+, CD23-, sIgM, cyclin D1 nuclear positivity is desirable but not essential
  * Central review of histology will be performed on diagnostic material
  * Molecular or cytogenetic confirmation of diagnosis is not required
* Previously untreated disease at any stage requiring therapy in the opinion of the treating physician

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 3 months

  * Life expectancy not severely limited by other illness
* Creatinine clearance ≥ 30 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study therapy
* No known serological positivity for HBV, HCV, or HIV
* No concurrent uncontrolled serious medical conditions
* No severe impairment of renal or liver function (alkaline phosphatase, bilirubin or creatinine > 2.5 times upper limit of normal) not related to lymphoma
* No known hypersensitivity to murine proteins
* No prior malignancy in the past 5 years, except for nonmelanoma skin tumor or curatively resected carcinoma in situ of the uterine cervix
* No history of a psychological illness or condition that, in the opinion of the investigator, may adversely affect compliance with study medication

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2006-12-07 (Actual); Primary Completion 2011-11-23 (Actual); Study Completion 2015-05-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of first administration of treatment until the date of death from any cause, assessed up to a maximum of 60 months
  Overall survival - Time from date of first administration of treatment until death from any cause

SECONDARY OUTCOMES:
Progression-free survival | From date of first treatment administration until the date of first documented progression or relapse, whichever came first, assessed up to a maximum of 60 months
  Progression-free survival - Time from date of first administration of treatment to Disease Progression or replapse
Toxicity - Number of patients with >=grade 3 toxicity | Within 30 days after last dose of treatment
  Toxicity - Number of patients who suffer grade 3 or 4 toxicities
Toxicity - Percentage of patients with >=grade 3 toxicity | Within 30 days after last dose of treatment
  Toxicity - Percentage of patients who suffer grade 3 or 4 toxicities
Tumor response duration | From date of first documentation of PR or CR until the date of first progression up to a maximum of 60 months
  Tumor response duration - Time from Complete or Partial Response to disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rule, MD, Principal Investigator — Derriford Hospital
Locations (67):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia
- United Kingdom (66):
  - William Harvey Hospital, Ashford, England
  - Stoke Mandeville Hospital, Aylesbury, England
  - Basingstoke and North Hampshire NHS Foundation Trust, Basingstoke, England
  - Royal United Hospital, Bath, England
  - Good Hope Hospital, Birmingham, England
  - Birmingham Heartlands Hospital, Birmingham, England
  - Blackpool Victoria Hospital, Blackpool, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - St. Helier Hospital, Carshalton, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Saint Richards Hospital, Chichester, England
  - Essex County Hospital, Colchester, England
  - Colchester General Hospital, Colchester, England
  - Queen Alexandra Hospital, Cosham, England
  - Mayday University Hospital, Croydon, England
  - Darlington Memorial, Darlington, England
  - Darent Valley Hospital, Dartford, England
  - Dewsbury and District Hospital, Dewsbury, England
  - Russells Hall Hospital, Dudley, England
  - Bishop Auckland Hospital, Durham, England
  - Epsom General Hospital, Epsom, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Medway Maritime Hospital, Gillingham, England
  - Gloucestershire Royal Hospital, Gloucester, England
  - Hereford Hospitals, Hereford, England
  - Wycombe General Hospital, High Wycombe, England
  - Leeds General Infirmary, Leeds, England
  - Cancer Research UK Clinical Centre at St. James's University Hospital, Leeds, England
  - Saint Bartholomew's Hospital, London, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Manchester Royal Infirmary, Manchester, England
  - Christie Hospital, Manchester, England
  - Queen Elizabeth The Queen Mother Hospital, Margate, England
  - Newcastle Upon Tyne Hospitals NHS Trust, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Norfolk and Norwich University Hospital, Norwich, England
  - Derriford Hospital, Plymouth, England
  - Pontefract General Infirmary, Pontefract, England
  - Portsmouth Oncology Centre at St Mary's Hospital, Portsmouth, England
  - Whiston Hospital, Prescot, England
  - Rosemere Cancer Centre at Royal Preston Hospital, Preston, England
  - East Surrey Hospital, Redhill, England
  - Pembury Hospital, Royal Tunbridge Wells, England
  - Kent and Sussex Hospital, Royal Tunbridge Wells, England
  - Salisbury District Hospital, Salisbury, England
  - Royal Hallamshire Hospital, Sheffield, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal South Hants Hospital, Southampton, England
  - Southampton General Hospital, Southampton, England
  - Sunderland Royal Hospital, Sunderland, England
  - Royal Marsden - Surrey, Sutton, England
  - Great Western Hospital, Swindon, England
  - Torbay Hospital, Torquay, England
  - Royal Cornwall Hospital, Truro, England
  - New Cross Hospital, Wolverhampton, England
  - Yeovil District Hospital, Yeovil, England
  - Monklands General Hospital, Airdrie, Scotland
  - Hairmyres Hospital, East Kilbride, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Pinderfields General Hospital, Wakefield, Scotland
  - Wishaw General Hospital, Wishaw, Scotland
  - Ysbyty Gwynedd, Bangor, Wales
  - Amersham Hospital, Amersham
  - Musgrove Park Hospital, Taunton

REFERENCES:
- [Derived] Rule S, Smith P, Johnson PW, Bolam S, Follows G, Gambell J, Hillmen P, Jack A, Johnson S, Kirkwood AA, Kruger A, Pocock C, Seymour JF, Toncheva M, Walewski J, Linch D. The addition of rituximab to fludarabine and cyclophosphamide chemotherapy results in a significant improvement in overall survival in patients with newly diagnosed mantle cell lymphoma: results of a randomized UK National Cancer Research Institute trial. Haematologica. 2016 Feb;101(2):235-40. doi: 10.3324/haematol.2015.128710. Epub 2015 Nov 26. PMID 26611473
- See also: Abstract on Pubmed — https://www.ncbi.nlm.nih.gov/pubmed/26611473
- See also: Publication in haematologica — http://www.haematologica.org/content/101/2/235.article-info